CLINICAL TRIAL: NCT02453867
Title: Multicenter, Prospective, Randomized Study Investigating the Efficacy and Safety of a Reduced Immunosuppressive Therapy With Tacrolimus Once Daily in Comparison to Standard Triple Immunosuppression in Senior Renal Transplant Recipients
Brief Title: Efficacy and Safety of a Reduced Immunosuppression vs. Standard Triple Therapy in Senior Renal Transplant Recipients
Acronym: REDUCE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klemens Budde (Other)
Collaborators: Charite University, Berlin, Germany (Other); European Renal Association - European Dialysis and Transplant Association (Other); European Kidney Transplant Association (EKITA) (Other); DESCARTES Working Group On Transplantation (Other)
Responsible Party: Sponsor-Investigator, Klemens Budde, Prof. Dr., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDUCE; 2014-002643-18 (EudraCT Number)
Record Dates: First submitted 2015-04-03; First posted 2015-05-27 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Immunosuppression After Renal Transplantation
Keywords: kidney transplantation; senior kidney transplant recipients; tacrolimus once daily; reduced immunosuppression; recipients >65 years; Senior
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard immunosuppression (Active Comparator): starting immunosuppression: tacrolimus (Advagraf) (target trough levels >5 ng/ml), mycophenolate mofetil >1g/d in MMF or >720 mg/d in mycophenolic acid, steroids from month 1-3 dosing according to local practice; 200 pts are planned to carry on with standard immunosuppression (tacrolimus (Advagraf), Mycophenolate, steroids) as stated above according to international guidelines for kidney transplant recipients from month 3 posttransplant to month 12 posttransplant
  Interventions: Drug: Tacrolimus; Drug: mycophenolate; Drug: Steroids
- Reduced immunosuppression (Experimental): The Intervention is stopping medication:
  200 pts are planned to receive a reduced immunosuppression after month 3: carry on with tacrolimus (Advagraf; trough levels >5 ng/ml) steroids stop at month 3 mycophenolate stop at month 6
  Interventions: Other: Reduced immunosuppression; Drug: Tacrolimus; Drug: mycophenolate

INTERVENTIONS:
Other: Reduced immunosuppression — Stop steroids at month 3 Stop mycophenolate at month 6 continue tacrolimus once daily (Advagraf, trough levels > 5ng/ml) Stop mycophenolate at month 6
  Arms: Reduced immunosuppression
Drug: Tacrolimus — Tacrolimus is used in both the acitve comparator arm and the interventional arm
  Other Names: Advagraf
Drug: mycophenolate — Mycophenolate is used in the acitve comparator arm for the whole study period; Mycophenolate is stopped at month 6 after Transplantation (month 3 of the study) in the experimental arm
Drug: Steroids — Steroids are used continually in the active comparator arm and are stopped at the beginning of the study (month 3 after Transplantation) as an Intervention in the experimental arm
  Arms: Standard immunosuppression

SUMMARY:
Study purpose To establish efficacy and safety of a reduced immunosuppressive therapy with tacrolimus once daily for senior (>65 years of age) renal transplant recipients

DETAILED DESCRIPTION:
Study outline Stable senior transplant recipients (>65 years of age) participating in the European SENIOR transplant registry may enter the trial at month 3 post-transplant, if they fulfil all of the in- and none of the exclusion criteria. At this time patients will be randomized 1:1 either to continue

Reference therapy:

Tacrolimus once daily (Advagraf®) Mycophenolate (either MMF ≥1g/d or EC-MPS ≥720g/d) Steroids (≥5mg prednisolone or equivalent) or to Investigational therapy: Tacrolimus once daily (Advagraf®) Steroid stop at month 3 (tapering within 2 weeks) Mycophenolate stop at month 6

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥65 years and participating in the European SENIOR transplant registry
2. Patients who received a renal allograft 3 - 3.5 months prior to randomization.
3. Patient must have received primary or secondary renal allograft from a blood group compatible donor
4. Standard criteria donors (SCD), expanded criteria donors (ECD), donors after cardiac death (DCD) and living donors (LD) are eligible
5. Patients who are willing and able to participate in the study and from whom written informed consent has been obtained
6. Patients on continuous standard triple therapy with tacrolimus once daily (Advagraf, trough level ≥5ng/ml) in combination with mycophenolate (either ≥1.0g/day MMF or ≥720mg/d EC-MPS) and steroids (≥5mg prednisolone or equivalent) since transplantation
7. Stable graft function with serum creatinine ≤2.5 mg/dl.
8. Patients with low to standard immunological risk, who had a PRA over 20% and no known donor specific antibodies (DSA) at transplantation

Exclusion Criteria:

1. Patient with mental dysfunction or inability to comply with the study protocol
2. Patients, who - according to the investigator - require for medical reasons (e.g. previous rejections) continuous triple therapy or a different tacrolimus exposure
3. Multi-organ recipients (other solid organ (e.g. pancreas) or bone marrow)
4. Blood group ABO-incompatible allografts
5. Patients who suffered from severe T-cell mediated rejection (over Banff II acute rejection), recurrent acute rejection (>1 episode), or steroid resistant rejection post-transplant
6. History of antibody-mediated rejection (acute or chronic)
7. History of rejection 2 months prior to inclusion
8. Documented presence of donor specific antibodies (DSA) according to local lab results at baseline
9. Panel reactive antibody (PRA) >20% prior to transplantation, measured according to local standard
10. Patients receiving or having received Sirolimus, Everolimus, Azathioprine, Belatacept or Cyclophosphamide within 3 months prior to enrolment
11. Patients having received any other induction therapy than Basiliximab (e.g. depleting polyclonal antithymocyte antibodies (ATG), OKT3, Alemtuzumab)
12. Patients with proteinuria >1.0 g/day (or >1.0 g/g creatinine) at screening or having experienced nephrotic syndrome due to recurrence of focal segmental glomerulosclerosis (FSGS)
13. History of alcohol or drug abuse with less than 6 months of sobriety
14. Patient with a known hereditary immunodeficiency
15. Patient with active malignancy posttransplant with the exception of local, non-invasive, fully excised, cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or cervical carcinoma in situ
16. Patients with clinically symptomatic congestive heart failure or symptomatic coronary artery disease
17. Patients with documented (either by serology and/or nuclear acid testing (NAT) clinically active infections (e.g. with a known Hepatitis B, Hepatitis C, HIV, CMV or BK virus infection)
18. Participation in any other investigational clinical trial 3 months before participation in this study, except the SENIOR transplant registry
19. Patients with leukopenia (<2500 cells/nl) or neutropenia (<1500 cells/nl)
20. Patients with thrombocytopenia (<100 cells/nl)
21. Patients with liver transaminases or bilirubin values > 3x normal values
22. Any significant diseases or clinically significant findings, including psychiatric and behavioural problems, medical history and/or physical examination findings that would in the opinion of the investigator preclude the patient from participating in the study.
23. Patients who have been institutionalized by official or court order

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Combined efficacy endpoint (BPAR, graft loss and death) | between randomization and month 12 posttransplant (month 9 of the study)
  BPAR (biopsy proven acute rejection)

SECONDARY OUTCOMES:
Number of severe infections | between randomization and month 12 posttransplant
  Numbers, type of infections will be registered
Number of opportunistic infections | between randomization and month 12 posttransplant
  CMV infections, BKV infections; numbers, type of infection will be registered
Number of hospitalisations and days of hospitalisation | between randomization and month 12 posttransplant
  number of episodes, days in hospital
Graft function by calculated glomarular filtration rate calculated by CKD-EPI | between randomization and month 12 posttransplant
  Comparison of estimated glomerular filtration rate calculated by CKD-EPI formula
Number of occurrences and types of donor specific antibodies (DSA) | between randomization and month 12 posttransplant
  surveillance of detection of new donor specific antibodies by Luminex assay

CONTACTS AND LOCATIONS:
Overall Officials: Klemens Budde, MD, Principal Investigator — Charite Universitaetsmedizin Berlin

IPD SHARING:
Plan to Share IPD: Yes
aggregated data are available through the Steering committee of DESCARTES and EKITA